CLINICAL TRIAL: NCT02299245
Title: Different Doses Rosuvastatin Effect on Telomere-telomerase System in Acute Coronary Syndrome Patients After Percutaneous Coronary INtervention: RETAIN Study
Brief Title: Rosuvastatin Effect on Telomere-telomerase System in ACS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Xiao-dong Zhuang (Other)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Sponsor-Investigator, Xiao-dong Zhuang, director of the department of cardiology, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RETAIN Study
Record Dates: First submitted 2014-11-14; First posted 2014-11-24 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2015-07

CONDITIONS: Telomere Shortening; Telomere Length, Mean Leukocyte; 22q Telomere Deletion Syndrome
Keywords: telomere; telomerase; statin; percutaneous coronary intervention; acute coronary syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- randomised to rosuvastatin (20mg/d) (Experimental): randomised to rosuvastatin (20mg/d)
  Interventions: Drug: rosuvastatin
- randomised to rosuvastatin (10mg/d) (Active Comparator): randomised to rosuvastatin (10mg/d)
  Interventions: Drug: rosuvastatin

INTERVENTIONS:
Drug: rosuvastatin — different dose of rosuvastatin treatment
  Other Names: Crestor

SUMMARY:
Coronary heart disease (CHD) is one of the diseases characterised by biological aging as one of the important risk factors in several epidemiological studies. The mean telomere length and telomerase activity serve as markers for the biological age at the cellular level, with shorter telomeres and lower telomerase activity defining the increased biological age. Telomere length and telomerase activity, therefore, correlates with the risk of CHD and atherosclerosis. A present study states that the treatment with a statin is associated with a reduction in the number of clinical events but only in individuals with increased risk based on their telomere length. This suggests a positive relationship of telomere and telomerase system with the treatment with statins in CHD patients.

DETAILED DESCRIPTION:
Coronary heart disease (CHD) is identified as one of the diseases characterised by biological aging as one of the important risk factors in several epidemiological studies. Premature biological aging is distinct from chronological aging and may predispose the individual to myocardial infarction, atherosclerosis and CHD in particular. The mean telomere length and telomerase activity serve as markers for the biological age at the cellular level, with shorter telomeres and lower telomerase activity defining the increased biological age. Telomere length and telomerase activity, therefore, correlates with the risk of CHD and atherosclerosis. Statins serve as the drugs of obvious choice based on their well established efficacy and safety profiles for the treatment of CHD and associated atherosclerosis. A present clinical study states that the treatment with a statin is associated with a reduction in the number of clinical events but only in individuals with increased risk based on their telomere length. This suggests a positive relationship of telomere and telomerase system with the risk of CHD and, therefore, would help clinicians to categorise the patient populations based on their leucocyte telomere length for treatment with statins.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with ACS, planing for PCI treatment
* Male or females who are 18-80years of age
* No current or previous statin therapy
* No current indication for statin therapy (Coronary artery disease; hypercholesterolemia, renal dysfunction)
* Subjects who have given their signed consent to participate in the study

Exclusion Criteria:

* Patient < 18 or > 80 years
* Renal dysfunction
* Hyperlipidemia
* Active myositis
* All forms of liver disease
* Pregnancy
* Breastfeeding
* Patients being treated with other type statin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-07 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in telomere length after different dose statin treatment | baseline; 4 and 24 weeks
  telomere length of circulating leukocyte will be measured by Southern blot test before and after treatment

SECONDARY OUTCOMES:
Change from baseline in telomerase activity after different dose statin treatment | baseline; 4 and 24 weeks
  telomerase activity of circulating leukocyte will be measured by Southern blot test before and after treatment
PCI-related myocardial infarction (MI) | PCI-related MI will be assesed within 24 hours after the end of the coronary artery stenting procedure
  PCI related myocardial infarction is defined by the third Universal definition of myocardial infarction